CLINICAL TRIAL: NCT06767540
Title: A Randomized Double-blind, Placebo-controlled, Multicenter Phase III Clinical Study Evaluating the Efficacy and Safety of AK120 in the Treatment of Moderate-to-severe Atopic Dermatitis (AD) in Adolescents
Brief Title: A Clinical Study of AK120 in Adolescents With Moderate-to-severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK120-302
Record Dates: First submitted 2025-01-08; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK120 600mg every two weeks (Q2W) subcutaneous injection (Experimental): AK120 600mg at day 1, then 300mg subcutaneous injection Q2W thereafter until week 46.
  Interventions: Drug: Placebo
- AK120 600mg every three weeks (Q3W) subcutaneous injection (Experimental): AK120 600mg at day 1, then 300mg subcutaneous injection Q3W thereafter until week 45.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Placebo — placebo subcutaneous injection Q2W until week 46.
  Arms: AK120 600mg every two weeks (Q2W) subcutaneous injection
Drug: placebo — placebo subcutaneous injection Q3W until week 45.
  Arms: AK120 600mg every three weeks (Q3W) subcutaneous injection

SUMMARY:
This is a randomized double-blind, placebo-controlled, multicenter phase III clinical study evaluating the efficacy and safety of AK120 in the treatment of moderate-to-severe AD in adolescents.

DETAILED DESCRIPTION:
This is a randomized double-blind, placebo-controlled, multicenter phase III clinical study to evaluate the safety and efficacy of AK120 in the treatment of moderate-to-severe AD in adolescents. The total duration of the study planned is approximately 57 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥12<18 years old, weight ≥ 30kg.
* AD diagnosed at least half a year before screening.
* Subject with EASI score ≥16, IGA ≥ 3, BSA ≥ 10% at screening and baseline
* Daily peak P-NRS scores (weekly average) at baseline visit ≥ 4.

Exclusion Criteria:

* Acute onset of AD in 4 weeks prior to enrollment.
* Undergone or planned surgery during the study period within the 4 weeks prior to enrollment, or unable to fully recover from surgery before enrollment.
* Previously suffered from vernal keratoconjunctivitis (VKC) or atopic keratoconjunctivitis (AKC).
* Received systemic traditional Chinese medicine treatment within the 4 weeks before randomization or topical traditional Chinese medicine treatment within 1 week before randomization.
* Received treatment with other clinical study drugs within 4 weeks or 5 halflives before randomization (whichever is longer).
* Have a history of allergies to any component of AK120 and/or severe allergic reactions to monoclonal antibodies.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-01-23 (Estimated); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who achieved Eczema Area and Severity Index (EASI)-75 | at week 18 （day 127)
  At week 18, the percentage of subjects who achieved EASI-75 compared to baseline. The EASI score ranges from 0 (no eczema) to 72 (maximum severity).
Percentage of subjects with the Investigator's Global Assessment (IGA) score decrease of ≥ 2 points | at week 18 （day 127)
  At week 18, the percentage of subjects with the IGA score decrease of ≥ 2 points from baseline. The IGA is a five-point scale ranging from 0 to 4 ( 0 indicates clear, 4 indicates severe).

SECONDARY OUTCOMES:
Percentage change in affected Body Surface Area (BSA) | week 0 to week 52
  Percentage change in BSA from baseline.
percentage change of Peak Pruritus Numerical Rating Scale (P-NRS) scores | week 0 to week 52
  percentage change of P-NRS scores from baseline at each visit. The scale ranging from 0 to 10 ( 0=no itch; 10=worst itch imaginable).
Percentage changes in the Children's Dermatology Life Quality Index (CDLQI) score | week 0 to week 52
  Percentage changes in the CDLQI score compared to baseline at each visit. The total score range from 0 to 30, with higher scores indicating a greater impact on the patient's quality of life.
Incidence of Adverse Events (AE) | week 0 to week 52
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - The Third People's Hospital of Zhuhai, Zhuhai, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Jinzhou Central Hospital, Jinzhou, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - XiangYa Hospital CentralSouth University, Changsha, Hunan
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Shandong Provincial Dermatology Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No